CLINICAL TRIAL: NCT06882395
Title: Impact of Aligner Replacement Protocols on Predictability of Planned Dental Movements: Evaluation of Double Aligner
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC.2024.Double_Aligner
Record Dates: First submitted 2025-03-07; First posted 2025-03-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-12

CONDITIONS: Malocclusion; Clear Aligner Appliance; Orthodontics; Tooth Movement
Keywords: Orthodontics; Tooth; Movement; Removable; Appliances
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: FLX aligner 10 days (Active Comparator): Participants use the FLX aligner exclusively for 10 days.
  Interventions: Device: Group 1: FLX aligners for 10 days
- Arm 2: FLX for 10 days + FLX35 for 3 days (Experimental): Participants use the FLX aligner for 7 days, followed by the FLX35 aligner for 3 days.
  Interventions: Device: Group 2: FLX aligners worn for 7 days, followed by FLX35 aligners for 3 days.
- FLX aligner for 7 days + FLX for 3 days (Experimental): FLX aligner for 7 days, followed by the FLX aligner for 3 days
  Interventions: Device: Group 3: FLX aligners for 7 days, followed by new FLX aligners for 3 days.

INTERVENTIONS:
Device: Group 1: FLX aligners for 10 days — FLX aligners worn for 10 days
  Arms: Arm 1: FLX aligner 10 days
Device: Group 3: FLX aligners for 7 days, followed by new FLX aligners for 3 days. — Group 3: FLX aligners worn for 7 days, followed by new FLX aligners for 3 days.
  Arms: FLX aligner for 7 days + FLX for 3 days
Device: Group 2: FLX aligners worn for 7 days, followed by FLX35 aligners for 3 days. — Group 2: FLX aligners for 7 days, followed by FLX35 aligners for 3 days.
  Arms: Arm 2: FLX for 10 days + FLX35 for 3 days

SUMMARY:
The study will evaluate the impact of replacing aligners after 7 days with new aligners made of different materials on the predictability of planned dental movements. Three groups of participants will follow different aligner protocols, and the planned movements will be compared with the achieved ones. The study aims to provide relevant data for clinical practices with orthodontic aligners and assess participants' satisfaction with the treatment.

DETAILED DESCRIPTION:
This prospective clinical trial aims to determine whether replacing an aligner after 7 days with a new aligner of a different material affects the predictability of planned dental movements. A total of 114 adult patients undergoing orthodontic treatment with aligners-requiring bilateral tooth movements (extrusion, intrusion, rotation, tipping, or mesiodistal translation)-will be recruited and randomized into three groups with distinct aligner exchange protocols.

Group 1: 10 days of exclusive FLX aligner use. Group 2: 7 days of FLX aligner use followed by 3 days of FLX35 use. Group 3: 7 days of FLX aligner use followed by 3 days of a new FLX aligner. Within each group, patients will be further categorized into subgroups based on horizontal, vertical, and rotational movements. Digital study models, radiographs, and standardized clinical photographs will be used to compare planned versus achieved tooth movements. The primary outcome is the predictability of movement, defined as the difference and percentage of planned versus actual movement. Secondary outcomes include participant satisfaction measured via the OHIP-14 questionnaire. Data will be analyzed using descriptive statistics and paired tests appropriate for the split-mouth design. The study is conducted in accordance with the Declaration of Helsinki, and all treatment costs will be covered by the sponsor, NeoDent (JJGC Industria e Comercio de Materiais Dentarios S.A.).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older, with full permanent dentition.
* Interested in orthodontic treatment with aligners.
* Planned movements include extrusion, intrusion, rotation, tipping, or mesiodistal translation.
* Signed informed consent.

Exclusion Criteria:

* Contraindications to aligner use, including allergies to polyurethane or PETG.
* Poor oral hygiene or active periodontal disease.
* Malocclusions involving multiple missing teeth or short clinical crowns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Tooth movement and predictability achieved by different aligner materials, evaluated through radiographs and intraoral scanning | 7 days
  Digital study models (obtained using an intraoral scanner), along with standardized digital panoramic and periapical radiographs, will be collected at three key stages: before treatment initiation (for diagnosis and planning), during treatment, and immediately after treatment completion (for assessing the results). This follows the standard clinical practice in orthodontic treatment.
  The intraoral scans will be analyzed in conjunction with the planned movement models generated by the orthodontic treatment planning software.
  To evaluate treatment efficacy, tooth tracking will be performed using Geomagic Control X. This analysis will compare the planned tooth movement (reported in mm) with the actual movement achieved (reported in mm). The planned movement aligns with the expected total. Therefore, the percentage (%) of orthodontic movement successfully completed will be calculated based on the measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Private orthodontic clinic, Curitba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No